CLINICAL TRIAL: NCT01815827
Title: An Open-label, Parallel Group Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of Inclacumab in Japanese Healthy Volunteers Compared to Caucasian Healthy Volunteers
Brief Title: A Study of Single Dose Inclacumab in Japanese Healthy Volunteers Compared to Caucasian Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: BP28134
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — inclacumab

ARMS (2):
- Caucasian Healthy volunteers (Active Comparator)
  Interventions: Drug: inclacumab
- Japanese Healthy volunteers (Experimental)
  Interventions: Drug: inclacumab

INTERVENTIONS:
Drug: inclacumab — single intravenous doses

SUMMARY:
This open-label, parallel group study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single doses of inclacumab in Japanese healthy volunteers compared to Caucasian healthy volunteers. Subjects will receive a single intravenous dose of inclacumab. Follow-up will be for up to 197 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, 18 to 55 years of age, inclusive Healthy status as defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history and a complete physical examination
* Japanese subjects must have Japanese parents and grandparents who were born in Japan
* Caucasian subjects must have Caucasian parents and grandparents
* Body mass index (BMI) 18 - 30 kg/m2 inclusive

Exclusion Criteria:

* Clinically significant abnormalities in laboratory test results (including positive test for HIV, hepatitis B and/or C), vital signs or ECGs
* Any confirmed significant allergic reactions against any drug, or multiple allergies (non-active hay fever is acceptable)
* Smokes more than 5 cigarettes per day during the three months prior to study conduct
* Participation in an investigational drug or device study within 30 days or 5 half-lives prior to screening
* Positive test for drugs of abuse
* Any suspicion of or history of alcohol and/or other substance abuse or addiction
* Pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve (AUC) | up to 197 days
Pharmacokinetics: Maximum plasma concentration (Cmax) | up to 197 days

SECONDARY OUTCOMES:
Pharmacodynamics: Blood platelet leukocytes aggregation (PLA) | up to 197 days
Pharmacodynamics: Plasma (free and total) soluble P-selectin | up to 197 days
Safety: Incidence of adverse events | approximately 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Anaheim, California, United States

REFERENCES:
- [Derived] Morrison M, Palermo G, Schmitt C. Lack of ethnic differences in the pharmacokinetics and pharmacodynamics of inclacumab in healthy Japanese and Caucasian subjects. Eur J Clin Pharmacol. 2015 Nov;71(11):1365-74. doi: 10.1007/s00228-015-1938-4. Epub 2015 Sep 12. PMID 26363899